CLINICAL TRIAL: NCT04562038
Title: Implementation of Electronic Shared Decision-Making Support for Families to Design and Monitor Participation-Focused Early Intervention
Brief Title: Implementation of Electronic Shared Decision-Making Support for Early Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Rocky Mountain Human Services (Other); University of Colorado, Denver (Other); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Mary A Khetani, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020-0555; AOTFIR20KHETANI (Other Grant/Funding Number: American Occupational Therapy Foundation)
Record Dates: First submitted 2020-07-19; First posted 2020-09-24 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Child Development Disorder; Development Delay
Keywords: early intervention; participation; shared decision-making; electronic; family-centered care
MeSH Terms: conditions — Developmental Disabilities; Learning Disabilities

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YC-PEM e-PRO (Experimental): Participants are administered an electronic patient-reported outcome measure to obtain information about parent priorities, and they obtain a summary report of their responses to share with their early intervention team for discussion during the annual IFSP meeting.
  Interventions: Behavioral: Young Children's Participation and Environment Measure (YC-PEM) electronic patient-reported outcome (e-PRO)
- Family Assessment (No Intervention): Participants are scheduled to complete a semi-structured family interview to obtain information about parent priorities, for use during the annual IFSP meeting

INTERVENTIONS:
Behavioral: Young Children's Participation and Environment Measure (YC-PEM) electronic patient-reported outcome (e-PRO) — The Young Children's Participation in Environment Measure (YC-PEM) is an evidence-based option for comprehensive proxy assessment of a young child's current and desired participation in occupations across home, daycare, and community settings. The YC-PEM is an electronic patient-reported outcome (e-PRO) that provides individual caregivers a valid, reliable, and feasible way to communicate information about their child's current participation in home and community activities and areas of participation need. The gained information is then summarized and shared with the child's EI provide team to identify intervention priorities and goal attainment strategies in partnership with families. For quality improvement, EI programs can aggregate the YC-PEM e-PRO data to examine trends in participation as a function of EI service use. It is therefore a promising electronic health systems intervention to enhance the parent-practitioner relationship, and an NIH common data element for trials.
  Arms: YC-PEM e-PRO

SUMMARY:
Family-centered care is a best practice approach to delivering high quality early intervention (EI) services for children 0-3 years old with developmental needs. Yet, family engagement in designing and monitoring their child's EI service plan is suboptimal. Families need a valid, reliable, and useful tool to share in decisions about the scope of their child's EI service plan. The investigators will achieve a major advance in contributing occupational therapy expertise to improve family engagement when designing and monitoring their child's EI services. The investigators will test the use of an evidence-based electronic tool with families at one EI program, when the child is due for an annual review of progress in the program. The investigators will also gather input from families, practitioners, and program leadership to identify facilitators and barriers to its use in multiple EI programs. This project tries to test an innovation in how the investigators deliver family-centered and participation-focused care. Study results will yield evidence for the effectiveness of the electronic intervention on parent activation, EI service plan focus, EI service use quantity, parent perceptions of EI service quality, and child functioning.

DETAILED DESCRIPTION:
Poor quality of care in early intervention (EI) is pervasive, particularly for vulnerable populations. Sub-optimal outcomes are perpetuated within this federally-funded, state administrated program due to significant cuts in federal per child appropriations. Optimizing EI outcomes will require ensuring the delivery of high value EI (i.e., providing services with the greatest reach, optimal outcomes, at the lowest cost). A lever to improve value-based EI is family-centered care, an evidence-based EI approach, which is grounded in family engagement and shared decision-making. Regrettably, the systematic implementation of strategies to empower families in this role are suboptimal, perpetuating poor outcomes and the failure of family-centered care. More than half of all EI enrolled families lack sufficient tools to engage in shared decision-making with EI practitioners when designing and monitoring the EI service plan. Therefore, if EI service quality and outcomes are going to be optimized, there is urgent need to equip families with a tool that will foster shared decision-making between the provider and family.

As EI programs transition to electronic data capture systems for accountability and quality improvement, the implementation of evidence-based electronic assessments is a scalable strategy to strengthen family engagement in shared decision-making to design and monitor EI services. One evidence-based option is the Young Children's Participation in Environment Measure (YC-PEM) electronic patient-reported outcome (e-PRO). The YC-PEM e-PRO has not been implemented into routine practice for families to communicate areas of participation difficulty for shared decision-making about intervention priorities.

The first aim is to conduct a community-based pragmatic trial of the Young Children's Participation and Environment Measure (YC-PEM), a valid electronic patient-reported outcome (e-PRO), at a single large, urban EI program to examine how this intervention is associated with: 1) EI service use breadth, intensity, and focus, 2) parent activation for shared decision making and engagement in EI services, 3) parent-reported EI service quality, and 3) gains in children's functioning.

EI service coordinators will be randomized to intervention and control groups arms, and then eligible and interested parents on their assigned caseloads will be assigned to the intervention and control groups as part of their child's annual evaluation of progress. Intervention group subjects will complete the YC-PEM e-PRO before the child's annual intervention planning meeting. EI service plan focus (participation-focused goals in the plan), EI service amount (breadth and intensity), EI service quality (parent-reported activation for shared decision-making to design EI services and parent satisfaction with family-centeredness of EI service delivery), and child functioning will be evaluated via electronic records and patient-reported outcomes data collected at baseline, and 4 weeks, 6 months, and 12 months.

AIM 1. Examine the effects of the YC-PEM e-PRO intervention on EI stakeholder outcomes.

(Aim 1a). Examine the effects of the YC-PEM e-PRO on EI parent activation, parent engagement in EI services, service plan focus, and service use breadth and intensity. The investigators will test two hypotheses in this first sub-aim. As compared to children receiving usual EI care, intervention group subjects will: H1: report higher activation for shared decision-making and parent engagement when planning and monitoring the child's EI care within 12 months; H2: receive a greater breadth and intensity of participation-focused EI services within 12 months.

(Aim 1b). Examine the effects of the YC-PEM e-PRO on parent report of EI service quality. As compared to usual care subjects, the investigators expect that parents in the intervention group will report greater satisfaction with: H1: enabling and partnership; H2: general and specific information exchange for shared decision-making; H3: coordinated and comprehensive EI care; and H4: respectful and supportive EI care.

(Aim 1c). Examine the effects of the YC-PEM e-PRO on child functioning. As compared to usual EI care, intervention group children will: H1: demonstrate greater developmental gains, as measured by state-mandated and norm-referenced developmental tests done at EI entry and 12 months. H2: demonstrate greater gains in functional skills, as measured by state-mandated outcomes data at EI entry and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver identifies as a parent or legal guardian of a child enrolled in early intervention
* Caregiver is at least 18 years old
* Caregiver reads, writes, and speaks English
* Caregiver has internet and telephone access
* Caregiver has a child who has received early intervention services for 3 or more months

Exclusion Criteria:

* Caregiver is not the parent or legal guardian of a child enrolled in early intervention
* Caregiver is 0-17 years old
* Caregiver does not read, write, or speak English
* Caregiver does not have internet or telephone access
* Caregiver does not have a child who has received early intervention services for 3 or more months

Ages: 3 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Measure of Processes of Care (MPOC-20) | Baseline (pre-intervention)
  Parent-reported EI quality; 20 items (7-point scale) assesses these domains of family-centered care: 1) enabling and partnership; 2) providing general and specific information; 3) coordinated and comprehensive care; and 4) respectful and supportive care.
Measure of Processes of Care (MPOC-20) | 4 weeks
  Parent-reported EI quality; 20 items (7-point scale) assesses these domains of family-centered care: 1) enabling and partnership; 2) providing general and specific information; 3) coordinated and comprehensive care; and 4) respectful and supportive care.
Measure of Processes of Care (MPOC-20) | 6 months
  Parent-reported EI quality; 20 items (7-point scale) assesses these domains of family-centered care: 1) enabling and partnership; 2) providing general and specific information; 3) coordinated and comprehensive care; and 4) respectful and supportive care.
Measure of Processes of Care (MPOC-20) | 12 months
  Parent-reported EI quality; 20 items (7-point scale) assesses these domains of family-centered care: 1) enabling and partnership; 2) providing general and specific information; 3) coordinated and comprehensive care; and 4) respectful and supportive care.

SECONDARY OUTCOMES:
Parent Patient Activation Measure (P-PAM) | Baseline (pre-intervention)
  Parent activation for shared decision-making; 13 items assesses parent knowledge, skills, and confidence to manage their child's care
Parent Patient Activation Measure (P-PAM) | 4 weeks
  Parent activation for shared decision-making; 13 items assesses parent knowledge, skills, and confidence to manage their child's care
Parent Patient Activation Measure (P-PAM) | 6 months
  Parent activation for shared decision-making; 13 items assesses parent knowledge, skills, and confidence to manage their child's care
Parent Patient Activation Measure (P-PAM) | 12 months
  Parent activation for shared decision-making; 13 items assesses parent knowledge, skills, and confidence to manage their child's care
Parent Participation Engagement measure (PPEM) | Baseline (pre-intervention)
  Parent engagement in EI services; 5 items (5-point scale) assesses parent active engagement in their child's EI services
Parent Participation Engagement measure (PPEM) | 4 weeks
  Parent engagement in EI services; 5 items (5-point scale) assesses parent active engagement in their child's EI services
Parent Participation Engagement measure (PPEM) | 6 months
  Parent engagement in EI services; 5 items (5-point scale) assesses parent active engagement in their child's EI services
Parent Participation Engagement measure (PPEM) | 12 months
  Parent engagement in EI services; 5 items (5-point scale) assesses parent active engagement in their child's EI services
Early Intervention Service Use Quantity | 1 month
  EI service use quantity will be captured according to service breadth and intensity. EI service breadth will be derived as a count of core EI services received (1, 2, 3+): physical therapy (PT), occupational therapy (OT), speech therapy (ST), developmental intervention (DI). For service intensity, estimates of service amount (hours) and service duration (months) from the service record will be used to derive an estimate of service use intensity (hours per month).
Early Intervention Service Use Quantity | 12 months
  EI service use quantity will be captured according to service breadth and intensity. EI service breadth will be derived as a count of core EI services received (1, 2, 3+): physical therapy (PT), occupational therapy (OT), speech therapy (ST), developmental intervention (DI). For service intensity, estimates of service amount (hours) and service duration (months) from the service record will be used to derive an estimate of service use intensity (hours per month).
Early Intervention Service Plan Focus | 4 weeks
  Record abstraction will be used to extract data on the child's service plan focus (i.e., EI service goals). These data will be coded using established quality criteria, to derive an estimate of the proportion of participation-focused goals in the EI service plan.
Child Functioning | Baseline (pre-intervention)
  Child Outcomes Summary (COS) scores that capture the child's functional capabilities. COS scores are a consensus rating by the EI team based on developmental scores and practitioner and parent perceptions of child function.
Child Functioning | 12 months
  Child Outcomes Summary (COS) scores that capture the child's functional capabilities. COS scores are a consensus rating by the EI team based on developmental scores and practitioner and parent perceptions of child function.

CONTACTS AND LOCATIONS:
Overall Officials: Mary A Khetani, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Rocky Mountain Human Services, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaelin V, Villegas V, Chen YF, Murphy N, Papautsky E, Litfin J, Leland N, Maheshwari V, McManus B, Khetani M; High Value Early Intervention Research Group. Effectiveness and scalability of an electronic patient-reported outcome measure and decision support tool for family-centred and participation-focused early intervention: PROSPECT hybrid type 1 trial protocol. BMJ Open. 2022 Jan 4;12(1):e051582. doi: 10.1136/bmjopen-2021-051582. PMID 34983760